CLINICAL TRIAL: NCT01775735
Title: Occipital Nerve Stimulation (ONS) for Migraine OPTIMISE
Brief Title: Occipital Nerve Stimulation (ONS) for Migraine: OPTIMISE
Acronym: OPTIMISE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: G120051; CDM00046436 (Other: BSC protocol number)
Record Dates: First submitted 2013-01-23; First posted 2013-01-25 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Migraine Disorders
Keywords: headache; pain; chronic
MeSH Terms: conditions — Migraine Disorders; Headache; Pain; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): The treatment is continuous stimulation with an occipital nerve stimulator, specifically the BSC Precision™ ONS System for 6 months post-randomization
  Interventions: Device: Occipital nerve stimulator
- Control (Active Comparator): The control is intermittent stimulation for 20 seconds every 90 minutes with an occipital nerve stimulator, specifically the BSC Precision™ ONS System for 6 months post-randomization
  Interventions: Device: Occipital nerve stimulator

INTERVENTIONS:
Device: Occipital nerve stimulator — Electrical stimulation of the greater occipital nerve
  Other Names: Boston Scientific Precision System

SUMMARY:
The primary objective of this study is to evaluate the safety and efficacy of occipital nerve stimulation (ONS) using the Boston Scientific Corporation (BSC) Precision™ System in the management of intractable chronic migraine, when used in conjunction with anti-migraine medications.

DETAILED DESCRIPTION:
Initial reports of managing migraine headache with ONS described a technique in which electrical leads were implanted in the subcutaneous space transverse to the occipital nerve, in the back of the head, under x-ray guidance. The leads were tunneled under the skin to an implantable pulse generator (IPG) implanted in the chest wall or abdomen. The OPTIMISE Trial is designed to be a pivotal study of the Boston Scientific PRECISION neurostimulation system, when the system is used for ONS. The PRECISION System has been previously been approved for Spinal Cord Stimulation (SCS).

ELIGIBILITY:
Key Inclusion Criteria:

* Onset of chronic migraine at least 6 months prior to start of Screening determined by a well-documented history
* Evidence of intractability
* Posterior-dominant head pain
* Stable pattern of headache symptoms for at least 6 months prior to the beginning of Screening
* Onset of migraine before the age of 50
* If female of childbearing potential: not pregnant, as evidenced by a negative pregnancy test

Key Exclusion Criteria:

* Diagnosed with any major psychiatric disorder not specifically listed in Key Exclusion Criteria 2-4 (e.g. multiple personality disorder, schizophrenia)
* Untreated panic disorder
* Untreated major depression evidenced by a PHQ-9 score >20
* Untreated generalized anxiety disorder evidenced by a GAD-7 score ≥15
* Currently diagnosed with severe personality disorder
* A female of childbearing potential planning to get pregnant during the course of the study or not using adequate contraception
* Participating in another drug, device, or biologics trial within 3 months prior to Screening
* A terminal illness associated with survival <24 months

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-04-10 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2017-01-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Lipton, MD, Principal Investigator — Albert Einstein College of Medicine
Locations (10):
- United States (10):
  - Boston Scientific Clinical Research Information Toll Free Number, Valencia, California
  - University of Illinois at Chicago (Implanting Physician), Chicago, Illinois
  - Diamond Headache Clinic (Headache Physician), Chicago, Illinois
  - Willis-Knighton River Cities Interventional Pain Specialist (Headache & Implanting Physician), Shreveport, Louisiana
  - Henry Ford Hospital (Headache Physician), Detroit, Michigan
  - Henry Ford Medical Group (Implanting Physician), West Bloomfield, Michigan
  - Mercy Pain Management -Surgery Center (Implanting Physician), Springfield, Missouri
  - Clinvest Research, LLC (Headache Physician), Springfield, Missouri
  - NYU Medical Center (Implanting Physician), New York, New York
  - Montefiore Headache Center (Headache Physician), The Bronx, New York

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 28 subjects were consented in the study. 13 failed screening and 15 were randomized. Statistically relevant conclusions cannot be made from this small sample size.
Period: Intervention (6 Months)
Arm/Group | Treatment | Control
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0
Period: Open Label (24 Months)
Arm/Group | Treatment | Control
Started | 8 | 7
Completed | 7 | 3
Not Completed | 1 | 4

BASELINE CHARACTERISTICS:
Population: Randomized subjects
Groups:
- Treatment: The treatment is continuous stimulation with an occipital nerve stimulator, specifically the BSC Precision™ ONS System
  Occipital nerve stimulator: Electrical stimulation of the greater occipital nerve
- Control: The control is intermittent stimulation for 20 seconds every 90 minutes with an occipital nerve stimulator, specifically the BSC Precision™ ONS System
  Occipital nerve stimulator: Electrical stimulation of the greater occipital nerve
- Total: Total of all reporting groups
Arm/Group | Treatment | Control | Total
Number analyzed (Participants) | 8 | 7 | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 7 | 14
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: American Indian or Alaska native | 0 | 0 | 0
  Race/Ethnicity: Asian | 0 | 0 | 0
  Race/Ethnicity: Black or African American | 0 | 0 | 0
  Race/Ethnicity: Hispanic or Latino | 1 | 0 | 1
  Race/Ethnicity: Native Hawaiian or other Pacific Islander | 0 | 0 | 0
  Race/Ethnicity: White | 7 | 7 | 14
  Race/Ethnicity: Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Moderate-to-severe Headache Days Per Month
Description: A moderate-to-severe headache day will be defined as any calendar day with:
  1. headache pain that lasts ≥4 hours AND peak severity of moderate or severe intensity
     OR
  2. a subject taking a triptan or ergot, regardless of headache pain duration or severity
  The Baseline number was calculated as the total count of eDiary calendar days which meet the definition of a moderate-to-severe headache day during the first 30 calendar days of eDiary entries if the eDiary contained ≥70% of data. The 6 months post-randomization number was calculated as the total count of eDiary calendar days which meet the definition of a moderate-to-severe headache day during the 30 calendar days of eDiary entries immediately preceding the subject's 6-Month Visit if the eDiary contained ≥70% of data.
Time Frame: from Baseline to 6 months post-randomization
Population: All subjects who completed Baseline and 6 months post-randomization and had ≥70% of eDiary data. Data for 5 subjects was not calculated due to missing eDiary data. Statistical analysis was not performed as the sample size is too small to draw any statistically relevant conclusions.
Measure: Median (Standard Deviation); unit: days
Arm/Group | Treatment | Control
Number analyzed (Participants) | 4 | 6
days | -5.2 (7.3) | 0 (10.8)

ADVERSE EVENTS:
Time Frame: Non-serious adverse events were collected from consent through the 6-month post-randomization visit. Serious adverse events were collected from consent through the 24-month post-randomization visit.
Arm/Group | Treatment | Control
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 4/8 | 1/7
Other Adverse Events (participants affected / at risk) | 3/8 | 3/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=8) | Control (N=7)
Migraine (Nervous system disorders) | 1 (12) | 0 (0)
Status migrainosus (Nervous system disorders) | 2 (2) | 0 (0)
Hemiplegic migraine (Nervous system disorders) | 1 (1) | 0 (0)
Migraine without aura (Nervous system disorders) | 1 (1) | 0 (0)
Adverse drug reaction (General disorders) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=8) | Control (N=7)
Implant site irritation (General disorders) | 1 (1) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Surgical skin tear (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed. Statistical analysis was not performed as the sample size was too small to draw any statistically relevant conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days